CLINICAL TRIAL: NCT00258310
Title: A Phase II Study Examining the Feasibility of Long Term and Low Dose Oral Capecitabine (Xeloda®) in Newly Diagnosed Head and Neck Squamous Cell Carcinoma (HNSCC) After Surgery, Radiation and/or Chemotherapy
Brief Title: Ph II Long Term/Low Dose Xeloda in Head and Neck Squamous Cell Carcinoma After Surgery, Radiation & or Chemo
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Barbara Ann Karmanos Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, George Yoo, Principal Investigator, Barbara Ann Karmanos Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2688; P30CA022453 (NIH); WSU-D-2688 (Other: Barbara Ann Karmanos Cancer Institute); WSU-HIC-120103M1F (Other: Wayne State University Institutional Review Board)
Record Dates: First submitted 2005-11-22; First posted 2005-11-24 (Estimated); Results first posted 2015-01-19 (Estimated); Last update posted 2023-03-10 (Actual); Status verified 2023-03

CONDITIONS: Head and Neck Cancer
Keywords: stage I squamous cell carcinoma of the hypopharynx; stage I squamous cell carcinoma of the larynx; stage I squamous cell carcinoma of the lip and oral cavity; stage I squamous cell carcinoma of the nasopharynx; stage I squamous cell carcinoma of the oropharynx; stage II squamous cell carcinoma of the hypopharynx; stage II squamous cell carcinoma of the larynx; stage II squamous cell carcinoma of the lip and oral cavity; stage II squamous cell carcinoma of the nasopharynx; stage II squamous cell carcinoma of the oropharynx; stage III squamous cell carcinoma of the hypopharynx; stage III squamous cell carcinoma of the larynx; stage III squamous cell carcinoma of the lip and oral cavity; stage III squamous cell carcinoma of the nasopharynx; stage III squamous cell carcinoma of the oropharynx; stage IV squamous cell carcinoma of the hypopharynx; stage IV squamous cell carcinoma of the larynx; stage IV squamous cell carcinoma of the lip and oral cavity; stage IV squamous cell carcinoma of the nasopharynx; stage IV squamous cell carcinoma of the oropharynx
MeSH Terms: conditions — Head and Neck Neoplasms; Squamous Cell Carcinoma of Head and Neck | interventions — Capecitabine; Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Capecitabine (Experimental): Surgery, chemotherapy and/or radiotherapy, prior to administration of Capecitabine 1000mg/day for one year.
  Interventions: Drug: capecitabine; Procedure: Surgery, chemotherapy and/or radiotherapy

INTERVENTIONS:
Drug: capecitabine — Capecitabine 1000mg/day for one year
  Other Names: Xeloda
Procedure: Surgery, chemotherapy and/or radiotherapy — Surgery, chemotherapy and/or radiotherapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as capecitabine, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving capecitabine after surgery, radiation therapy, and/or chemotherapy may kill any remaining tumor cells.

PURPOSE: This phase II trial is studying how well capecitabine works in treating patients who have undergone previous surgery, radiation therapy, and/or chemotherapy for head and neck cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the feasibility of adjuvant low-dose capecitabine in patients with squamous cell carcinoma of the head and neck who have undergone prior curative surgery, radiotherapy, and/or chemotherapy.

Secondary

* Determine the time to recurrence, local-regional control, and survival rate in patients treated with this drug.
* Determine the incidence of second primary tumors in patients treated with this drug.

OUTLINE: This is an open-label study.

Patients receive oral capecitabine once daily for 1 year in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed every 3 months for 1 year and then every 6 months for 1 year.

PROJECTED ACCRUAL: A total of 41 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed squamous cell carcinoma of the head and neck, including 1 of the following primary tumor sites:

  * Oral cavity
  * Oropharynx
  * Nasopharynx
  * Hypopharynx
  * Larynx
  * Unknown primary
* Any disease stage allowed
* No evidence of active disease
* Must have undergone curative surgical resection, radiotherapy, and/or chemotherapy at least 1 month, but no more than 4 years ago

PATIENT CHARACTERISTICS:

Performance status

* Karnofsky 70-100%

Life expectancy

* More than 3 months

Hematopoietic

* White blood count (WBC) ≥ 3,000/mm^3
* Granulocyte count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3

Hepatic

* Bilirubin ≤ 1.5 times upper limit of normal (ULN)
* Aspartate Aminotransferase (AST) or Alanine Aminotransferase (ALT) ≤ 2.5 times ULN
* Alkaline phosphatase ≤ 2.5 times ULN
* Hepatitis B and/or C negative

Renal

* Creatinine clearance > 50 mL/min

Cardiovascular

* No myocardial infarction within the past 12 months
* No uncontrolled congestive heart failure
* No unstable or uncontrolled angina

Gastrointestinal

* No lack of physical integrity of the upper gastrointestinal tract
* Must be able to swallow tablet
* No malabsorption syndrome

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* HIV negative
* No other malignancy within the past 5 years except adequately treated basal cell or squamous cell skin cancer, carcinoma in situ of the cervix, or stage I or II cancer for which the patient is currently in complete remission
* No history of uncontrolled seizures, central nervous system (CNS) disorders, or psychiatric disability that would preclude study compliance or giving informed consent
* No ongoing postoperative fistula
* No prior unanticipated severe reaction to fluoropyrimidine therapy or known sensitivity to fluorouracil
* No other serious uncontrolled medical or surgical condition that would preclude study participation

PRIOR CONCURRENT THERAPY:

Chemotherapy

* See Disease Characteristics
* Prior oral fluoropyrimidine therapy allowed provided it was given in the adjuvant setting and completed ≥ 12 months ago

Radiotherapy

* See Disease Characteristics

Surgery

* See Disease Characteristics
* More than 4 weeks since prior major surgery and recovered
* No prior organ allografts

Other

* More than 4 weeks since prior participation in any investigational drug study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2003-12; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: George H. Yoo, MD, Study Chair — Barbara Ann Karmanos Cancer Institute
Locations (1):
- Barbara Ann Karmanos Cancer Institute, Detroit, Michigan, United States

REFERENCES:
- See also: Clinical trial summary from the National Cancer Institute's PDQ® database — http://cancer.gov/clinicaltrials

RESULTS

PARTICIPANT FLOW:
Groups:
- Capecitabine: Capecitabine 1000mg/day for one year
  capecitabine
  adjuvant therapy
Period: Overall Study
Arm/Group | Capecitabine
Started | 35
Completed | 35
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Capecitabine
Number analyzed (Participants) | 35
Age, Continuous [Median (Full Range); unit: years] | 58 [43 to 74]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 28
Region of Enrollment [Number; unit: participants]
  United States | 35

OUTCOME MEASURES:

1. Primary Outcome: Compliance With Treatment .
Description: Compliance is defined as taking at least 80% of the prescribed dose for one year.
Time Frame: within 365 days
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Capecitabine
Number analyzed (Participants) | 35
percentage of participants | 74 [59 to 90]
Statistical Analysis 1: Comparison: Capecitabine; Test type: Superiority or Other; proportion = 0.74, 95% CI 2-sided [.59 to .90]

2. Secondary Outcome: Recurrence-free Survival
Description: Time to recurrence or death
Time Frame: Within 3 years of end of study.
Population: All enrolled participants
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Capecitabine
Number analyzed (Participants) | 34
months | NA [NA to NA] — Median was not reached due to insufficient number of participants with events

3. Secondary Outcome: Overall Survival
Description: Estimated time from study entry to death from any cause
Time Frame: Within 3 years of end of study
Population: Entire study population
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Capecitabine
Number analyzed (Participants) | 33
months | NA [NA to NA] — Neither the median nor the 95% confidence interval can be calculated because there were too few deaths.

4. Secondary Outcome: Incidence of Second Primary Tumors
Time Frame: Within 3 years of end of study
Population: Entire study population
Measure: Count of Participants; unit: Participants
Arm/Group | Capecitabine
Number analyzed (Participants) | 35
Participants | 3

ADVERSE EVENTS:
Groups:
- Capcitabine: Capecitabine 1000mg/day for one year
  adjuvant therapy
Arm/Group | Capcitabine
Serious Adverse Events (participants affected / at risk) | 2/35
Other Adverse Events (participants affected / at risk) | 3/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Capcitabine (N=35)
Respiratory Failure (Cardiac disorders) | 1 (1)
Hand Foot Syndrome (General disorders) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Capcitabine (N=35)
Nausea/vomiting (Gastrointestinal disorders) | 3 (3)

LIMITATIONS AND CAVEATS:
There were no significant limitations.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No